CLINICAL TRIAL: NCT03153904
Title: Child STEPs for Youth Mental Health in Connecticut
Brief Title: Connecticut Child STEPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, John Weisz, Professor and Primary Investigator, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-1904
Record Dates: First submitted 2017-03-28; First posted 2017-05-15 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Anxiety; Depression; Trauma; Behavior Problems
Keywords: anxiety; depression; trauma; behavior problems; evidence-based treatments; manualized treatments; cognitive-behavioral therapy; youth; mental health
MeSH Terms: conditions — Anxiety Disorders; Depression; Wounds and Injuries; Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MATCH Training plus MATCH Consultation (Experimental): Therapists at local, community clinics attend a 6-day training on the Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, and Conduct Problems (MATCH; Chorpita & Weisz, 2009). After the training, therapists participate in weekly consultation meetings that are led by a MATCH Consultant from the study team. MATCH Consultants review sessions and the clinical monitoring and feedback system, provide recommendations for upcoming sessions, and review MATCH modules via role-plays and models.
  Interventions: Behavioral: Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, and Conduct Problems; Other: Monitoring and Feedback System
- MATCH Training only (Active Comparator): Therapists at local, community clinics attend a 6-day training on the Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, and Conduct Problems (MATCH; Chorpita & Weisz, 2009). After the training, therapists use MATCH as they think best and receive supervision from supervisors at the clinic.
  Interventions: Behavioral: Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, and Conduct Problems; Other: Monitoring and Feedback System

INTERVENTIONS:
Behavioral: Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, and Conduct Problems — MATCH-ADTC (Chorpita & Weisz, 2009) is designed for children aged 6-15. Unlike most evidence-based treatments (EBTs), which focus on single disorder categories (e.g., anxiety only), MATCH is designed for multiple disorders and problems encompassing anxiety, depression, post-traumatic stress, and disruptive conduct, including the conduct problems associated with ADHD. MATCH is composed of 33 modules-i.e., specific treatment procedures derived from decades of research on EBTs. The various modules can be organized and sequenced flexibly to tailor treatment to each child's characteristics and needs.
  Other Names: MATCH; MATCH - ADTC
Other: Monitoring and Feedback System — For each child, the web-based MFS provides weekly monitoring of the MATCH modules used and the child's treatment response, in two forms (a) changes on the Brief Problem Monitor (BPM) and (b) changes in severity of the top treatment concerns identified by youths and caregivers. At the end of treatment, the MFS provides a complete record of modules used, and child treatment response, across all weeks of treatment.
  Other Names: MFS

SUMMARY:
Connecticut Child STEPS is a randomized controlled trail investigating the effectiveness of MATCH-ADTC in treating anxiety, depression, trauma, and/or behavioral problems in children seeking services at four Department of Children and Families (DCF) funded clinics in the state of Connecticut. The study will evaluate child outcomes following two forms of therapist training in the MATCH model.

DETAILED DESCRIPTION:
This randomized controlled trial (RCT) will investigate the effectiveness of a modular, transdiagnostic treatment protocol for youth with anxiety, depression, trauma, and/or behavioral problems (MATCH-ADTC) in four DCF funded clinics in the state of Connecticut. MATCH synthesizes common elements found across dozens of evidence-based treatments into one model that is flexible and responsive to the complex needs of children and families. The RCT will evaluate child outcomes following two forms of therapist training in the MATCH model: (1) the 6-day MATCH training only; (2) the 6-day MATCH training plus weekly ongoing case consultation with a MATCH consultant. Participating children are between the ages of 7 and 15.

ELIGIBILITY:
Inclusion Criteria:

1. 7 to 15 year old child and their caregivers
2. seeking services at community mental health clinics
3. primary problem or disorder related to anxiety, traumatic stress, depression, or conduct problems, or any combination of the four problems

Exclusion Criteria:

1. child is outside of 7-15 age range
2. child does not have elevations in the areas of anxiety, depression, conduct, or posttraumatic stress
3. child is experiencing other primary clinical problems outside of MATCH focus such as:

   * ADHD identified as primary reason for seeking treatment
   * Schizophrenic spectrum disorder including Major Depressive Disorder with psychotic features
   * Autism spectrum disorder including Pervasive Developmental Disorder, Asperger's Disorder, Child Disintegrative Disorder, Rett's Disorder
   * Eating disorder including Anorexia Nervosa and Bulimia Nervosa
   * Mental Retardation
4. having been hospitalized for suicidal thoughts or behaviors within the past year
5. if the problem area of focus is beyond the scope of outpatient treatment and MATCH (e.g., severe aggression, psychosis, severe current suicidal ideation)
6. if child does not have a primary caregiver that can be involved in treatment and complete research assessments

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2013-10; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Brief Problem Monitor (BPM) | Weekly from baseline to the end of treatment, and every three months therafter until 18 month follow-up
Top Problems Assessment (TPA) | Weekly from baseline to the end of treatment, and every three months therafter until 18 month follow-up

SECONDARY OUTCOMES:
Therapist Satisfaction Inventory (TSI) | Change over time from Day 1 to end of treatment, an average of 22 weeks after baseline
Youth Services Survey for Families (YSS-F) | Post-treatment, an average of 22 weeks after baseline
Youth Self-Report and Child Behavior Checklist | Change over time from Day 1 to 18 month follow-up
Evidence-Based Practice Attitudes Scale (EBPAS) | Post-treatment, an average of 22 weeks after baseline
Early Adolescent Temperament Questionnaire Revised (EATQ-R) | Change over time from Day 1 to 18 month follow-up
Child Satisfaction Survey (CSC) | Post-treatment, an average of 22 weeks after baseline
Therapeutic Alliance Scale for Children (TASC) | Post-treatment, an average of 22 weeks after baseline

CONTACTS AND LOCATIONS:
Overall Officials: John R Weisz, PhD, Principal Investigator — Harvard University
Locations (1):
- Harvard University, Cambridge, Massachusetts, United States

REFERENCES:
- [Background] Chorpita, B.F., & Weisz, J.R. (2009). Modular Approach to Therapy for Children with Anxiety, Depression, Trauma, or Conduct Problems (MATCH-ADTC). Satellite Beach, FL: PracticeWise, LLC.
- [Derived] Johansen K, Saran I, Cho E, Weisz JR, Price MA. Examining racial and ethnic differences in youth psychotherapy treatment engagement and outcomes. J Consult Clin Psychol. 2024 Nov;92(11):769-778. doi: 10.1037/ccp0000919. PMID 39621369
- [Derived] Susman ES, Weisz JR, McLaughlin KA, Coulombe P, Evans SC, Thomassin K. Is respiratory sinus arrhythmia a modifiable index of symptom change in cognitive behavioral therapy for youth? A pooled-data analysis of a randomized trial. Psychother Res. 2025 Feb;35(2):337-351. doi: 10.1080/10503307.2024.2308149. Epub 2024 Jan 29. PMID 38285175
- [Derived] Evans SC, Wei MA, Harmon SL, Weisz JR. Modular Psychotherapy Outcomes for Youth With Different Latent Profiles of Irritability and Emotion Dysregulation. Front Psychiatry. 2021 Apr 16;12:618455. doi: 10.3389/fpsyt.2021.618455. eCollection 2021. PMID 33935825
- [Derived] Weisz JR, Thomassin K, Hersh J, Santucci LC, MacPherson HA, Rodriguez GM, Bearman SK, Lang JM, Vanderploeg JJ, Marshall TM, Lu JJ, Jensen-Doss A, Evans SC. Clinician training, then what? Randomized clinical trial of child STEPs psychotherapy using lower-cost implementation supports with versus without expert consultation. J Consult Clin Psychol. 2020 Dec;88(12):1065-1078. doi: 10.1037/ccp0000536. PMID 33370131